CLINICAL TRIAL: NCT01808274
Title: Safety and Performance Study of the Edwards CENTERA Self-Expanding Transcatheter Heart Valve
Acronym: CENTERA-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Collaborators: Medstar Health Research Institute (Other); European Cardiovascular Research Center (Network); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-03
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Aortic Valve Disease
Keywords: Transcatheter Aortic Valve Replacement; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAVR (Experimental): with CENTERA self-expanding valve
  Interventions: Device: Edwards CENTERA Self-Expanding Transcatheter Heart Valve

INTERVENTIONS:
Device: Edwards CENTERA Self-Expanding Transcatheter Heart Valve — The Edwards CENTERA Transcatheter Heart Valve (THV) System is indicated for use in symptomatic patients (high surgical risk) with severe aortic stenosis requiring aortic valve replacement (AVR).
  Other Names: TAVR; TAVI

SUMMARY:
The purpose of this study is to assess the safety and device success of the Edwards CENTERA Transcatheter Heart Valve (THV) System in patients with symptomatic, severe aortic stenosis who are indicated for aortic valve replacement.

DETAILED DESCRIPTION:
This is a non-randomized, prospective, multi-center safety and device success study. 34 patients have been enrolled at 4 participating investigational centers in Europe. Patient participation will last for a minimum of 5 years. Patients will be assessed at the following intervals: baseline, discharge, 30 days, 6 months, 1 year and annually thereafter through 5 years

ELIGIBILITY:
Inclusion Criteria:

1. High surgical risk: STS Score ≥ 8,EuroSCORE ≥ 15.
2. NYHA ≥ II.
3. Heart team (including examining cardiac surgeon) agrees on eligibility including assessment that TAVR is appropriate.
4. Study patient is an adult of legal consent age.
5. Study patient has provided written informed consent to comply with all of the study procedures and follow-up visits.

Exclusion Criteria:

1. Acute myocardial infarction ≤ 30 days before the intended treatment.
2. Untreated clinically significant coronary artery disease requiring revascularization.
3. Aortic valve is a congenital unicuspid or congenital bicuspid valve.
4. Mixed aortic valve disease (with predominant aortic regurgitation).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2013-09-17 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
All-cause mortality rate | 30 days post-index procedure
  NAP

SECONDARY OUTCOMES:
device success | 30 days
  Device success is defined as a composite of the following events:
  Factor 1: Absence of procedural mortality Factor 2: Correct positioning of a single prosthetic valve into the proper anatomical location Factor 3: Intended performance of the prosthetic heart valve (per the 30-day core lab echo assessment).
  It is measured in % (favorable measures/total measures).
device success | 1 year
  Device success is defined as a composite of the following events:
  Factor 1: Absence of procedural mortality Factor 2: Correct positioning of a single prosthetic valve into the proper anatomical location Factor 3: Intended performance of the prosthetic heart valve (per the 30-day core lab echo assessment).
  It is measured in % (favorable measures/total measures).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Windecker, MD, Principal Investigator — Inselspital Bern (Switzerland); Prof. Mohr, MD, Principal Investigator — Leipzig, Rhön Herzentrum (Germany)
Locations (4):
- Germany (3):
  - Herzzentrum Universitaet Bonn, Bonn
  - Asklepios Klinik St Georg Hamburg, Hamburg
  - Heart Center Leipzig, Leipzig
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No